CLINICAL TRIAL: NCT05820594
Title: A Feasibility Study of Controlled Human Infection With Intradermal Bacillus Calmette-Guérin Injection
Brief Title: Using BCG Vaccine to Understand Tuberculosis Infection
Acronym: Pilot BCG CHIM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Liverpool School of Tropical Medicine (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 23-005; 321376 (Other: Integrated Research Application System (IRAS))
Record Dates: First submitted 2023-03-22; First posted 2023-04-19 (Actual); Last update posted 2023-07-07 (Actual); Status verified 2023-04

CONDITIONS: Tuberculosis
Keywords: BCG; bacille calmette-guérin; Human challenge; Controlled human infection
MeSH Terms: conditions — Tuberculosis | interventions — BCG Vaccine

STUDY DESIGN:
Intervention Model Description: Single centre, prospective longitudinal controlled human infection study after intradermal injection with BCG SSI
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intradermal injection with BCG SSI (Experimental): Intradermal injection with BCG (bacillus calmette-guerin) vaccine at day 0.
  Interventions: Biological: Intradermal BCG (bacillus calmette-guerin) vaccine AJV

INTERVENTIONS:
Biological: Intradermal BCG (bacillus calmette-guerin) vaccine AJV — Participants will receive a one off dose of BCG (bacillus calmette-guerin) Vaccine AJV which contains the Danish Strain of Mycobacterium bovis BCG at a dose of 6 - 24 x 105 CFU (three times the standard dose). This will be injected intradermally into the upper deltoid region.

SUMMARY:
Tuberculosis (TB) is a disease that usually causes an infection in the lungs. The only vaccine to prevent TB is called BCG (Bacillus Calmette-Guérin). BCG contains a live germ similar to Mycobacterium tuberculosis, the germ that causes TB. BCG does not work very well, and TB remains the most common cause of death by infection worldwide. Human challenge models involve exposing healthy volunteers to an infectious disease in a safe and controlled way. This helps researchers understand more about an infectious disease and the body's response and can help develop new vaccines and treatments. The purpose of this study is to set up a human challenge model using BCG to understand how the body responds to this. If our human challenge model works well it may be used to help researchers develop new vaccines and tablets to treat TB in the future.

This study will recruit healthy volunteers, of all genders, age 18-50 years. The first part of the study (phase A) will recruit 10 participants. Participants in phase A will receive intradermal injection with BCG into the upper arm at three times the usual dose. On day 14 after BCG the following skin samples will be taken from the BCG site with the use of local anaesthetic: skin swab, microbiopsy, skin scrape and punch biopsy. Participants in this phase of the study will also have blood tests to ensure they are safe to take part and to monitor the immune response to BCG. The overall aim of this part of the study will be to ensure BCG can be isolated (grown in culture and by molecular techniques) from participants' BCG site 14 days after the injection. The investigators aim to test whether BCG can be isolated by punch biopsy and minimally invasive techniques (microbiopsy, skin scrape and skin swab). If the investigators find that they can isolate BCG successfully using the minimally invasive methods of skin sampling and the participants have not experienced any serious adverse events, they can proceed to phase B of the study.

In phase B 20 participants will be recruited. These participants will receive BCG as described for phase A. They will then have serial skin samples taken using either microbiopsy, skin scrape or skin swab on days 0, 2, 7, 14 and 28. The focus of this phase of the study is to assess immune responses to intradermal injection at the local (skin), systemic (blood) and respiratory mucosal (nose) compartments. This will involve longitudinal sampling from blood, nose and skin to measure BCG growth and the immune response over time.

DETAILED DESCRIPTION:
Background In 2020 an estimated 10 million people fell ill with tuberculosis (TB) and 1.5 million people died making TB the second leading infectious killer after COVID-19. Multi-drug resistant tuberculosis is a public health crisis and increasing health security threat. Despite this, the only currently available vaccine for prevention of tuberculosis is the 100-year-old Bacille Calmette-Guerin (BCG), which prevents disseminated forms of tuberculosis but has limited efficacy against pulmonary tuberculosis.

Phase 3 vaccine trials for tuberculosis are large, costly and conducted over prolonged periods. Controlled human infection models involve inoculating healthy participants with an infectious agent and can be used to accelerate vaccine development as well as improve understanding of disease pathogenesis and the host immune response and the development of new therapeutic combinations. There are current concerns in using wild type Mycobacterium tuberculosis as a human challenge agent given that infection cannot be reliably eradicated. The McShane group in Oxford have established a human challenge model using intradermal BCG and have published several peer reviewed articles. The Liverpool School of Tropical Medicine propose to replicate and further refine this model and I will be undertaking this project as part of an MD. The investigators aim to perform serial skin sampling paired with respiratory mucosal and systemic sampling to investigate and compare the immune response between these compartments. Ultimately this model may be used to select the most promising candidates for clinical trials.

Study hypothesis

1. BCG SSI strain will be recovered by tissue biopsy 14 days after intradermal injection by both classical microbiological and molecular diagnostic techniques.
2. Quantified BCG recovery (molecular techniques) by minimally invasive skin biopsy will be at least 90% as good as gold standard punch biopsy and will offer a more acceptable method for participants in the future.

Overall study design This is a single-centre study divided into two parts. The first part of the study (phase A) will recruit 10 participants. The participants in phase A will receive intradermal injection of BCG SSI vaccine into the upper arm on day 0 at three times the usual dose (BCG SSI 6-24 x 105 colony forming units). On day 14 after BCG injection. the following skin samples will be taken from the BCG injection site with the use of local anaesthetic: skin swab, microbiopsy, skin scrape and punch biopsy. The overall aim of this part of the study will be to ensure BCG can be isolated from participants BCG intradermal injection site 14 days after the injection. The investigators aim to test whether BCG can be isolated in comparable amounts by punch biopsy and minimally invasive techniques (microbiopsy, skin scrape and skin swab). They will proceed to phase B of the study if they are able to isolate BCG by culture or PCR using one of the minimally invasive techniques and no serious adverse events have occurred.

In the second phase of the study (phase B) 20 participants will be recruited. These participants will receive the BCG vaccine as described for phase A. The minimally invasive technique with the best BCG recovery will be used to perform longitudinal skin sampling to monitor BCG growth and the local skin immune response. Parallel samples will be taken from the respiratory mucosa and blood to compare the immune response in these compartments.

Study procedures

Consent:

In both phases of the study the consent and screening process will be the same. Potential participants will be invited to discuss the study at a 60 minute appointment, where they will watch a presentation on the study and complete a consent quiz to demonstrate understanding of the study and capacity to consent.

Screening:

To assess eligibility for the study, a focused medical history will be taken. If deemed necessary by the research team, GP questionnaires will be sent to GPs of participants if their vaccination history or medical history is unclear. A clinical examination will be performed including cardiorespiratory examination. Vital signs will be taken, as well as a nose and throat swab for COVID-19 lateral flow test (if required by UKHSA) and storage, urine pregnancy test (females only). The following blood tests will be taken: HIV test, hepatitis serology, full blood count and clotting, stored serum, blood PBMCs.

BCG intradermal injection (day 0):

For both parts of the study, at the BCG injection visit, participants will receive a single injection of the BCG vaccine at three times the usual dose intradermally into the upper arm. A CE marked intradermal delivery device (NanoPass MicronJet, NanoPass Technologies Ltd) will be used, which is licensed for the intradermal delivery of liquid drugs including vaccines for standardised intradermal delivery. After this visit participants will complete an electronic diary for 14 days to report any adverse events. Throughout the study, participants will have access to a 24/7 on-call telephone service.

Follow-up phase A:

In phase A, participants will attend follow-up appointments on days 2, 7, 14, 21 and 28 after BCG. A skin swab will be taken from the BCG injection site and a photograph of the site at each follow-up visit. The following blood tests will be taken: serum and PBMC for immunology ate each follow up visit and blood RNA on day 2.

In addition participants will attend on day 14 for skin biopsies. Local anaesthetic will be injected around the BCG vaccination site and the following skin samples will be taken in this order:

* Microbiopsy - This instrument uses a hollow needle to take a skin sample of 0.21mm diameter, 0.4mm depth.
* Skin scrape - This will take a sample from the skin surface using a Rhino-probe.
* Punch biopsy - This will take a skin sample from the middle of the BCG site using a 4mm punch biopsy instrument.

Follow-up Phase B:

In phase B participants will attend for follow-up visits on days 2, 7, 14, 21 and 28 after the BCG injection as with phase A.

In addition, in phase B the following respiratory mucosal samples will be taken from the nose on days 0, 2, 7, 14, 21 and 28 in phase B:

* Nasal wash will be performed in a subset of participants only- the nose is irrigated with normal saline and the liquid that is produced is collected and analysed
* Nasosorption - participants will have small pieces of filter paper inserted into nostrils for maximum of 2 minutes
* Nasal scrape - small superficial scrapes are taken from inside the nose to collect nasal cells
* The following skin samples will be taken from the BCG vaccination site: Microbiopsy OR skin scrape (depending on results of phase A) AND Skin swab on days 0, 2, 7, 14, 21 and 28

Laboratory mycobacteriological analysis

* Skin biopsy specimens will be cryopreserved and subsequently processed in batch
* Skin samples will be thawed and homogenised then cultured on Middlebrook 7H11 agar for 4 weeks before counting.
* The remaining biopsy specimen homogenate will be stored at -80° for subsequent DNA extraction
* The remaining homegenate will be thawed and DNA will be extracted and quantitative PCR will be performed

Laboratory immunological analysis Antibody responses: Samples of serum and nasosorption will be retained for antibody measurement using standard ELISA assays.

Cellular responses: Ex Vivo Interferon γ (IFN-γ) Enzyme-Linked Immunospot (ELISpot) assays will be performed on freshly isolated PBMCs from all participants. Responses to purified protein derivative (PPD) from M. tuberculosis will also be assessed. Unstimulated PBMCs will be used as a measure of background IFN-γ production. Results will be reported as spot-forming cells per million PBMCs, calculated by subtracting the mean count of the unstimulated PBMCs from the mean count of triplicate antigen wells and correcting for number of PBMCs in the well.

RNA analysis: Samples will be retained for transcriptomic signature feasibility testing. These methods will be essential as the CHIM develops for vaccine testing.

Reporting procedures for serious adverse events (SAEs) and suspected unexpected serious adverse reactions (SUSARs):

Adverse events will be actively and passively solicited. A symptom diary will be completed for the first 14 days to identify any adverse events and adverse events will be solicited at follow-up visits and recorded in the participant eCRF. Any serious adverse event considered by the CI to be related to the challenge agent and unexpected will be reported to the REC. As the challenge agents are vaccines with Marketing Authorisation, the mechanism for reporting any SAEs to the MHRA is via yellow card.

Data and Safety Monitoring Committee (DSMC)

The specific role of the committee will be:

* To independently review SAEs and AESIs regardless of relatedness to any of the study procedures throughout the study.
* To formally review the safety profile and quantified BCG recovery rate
* To perform unscheduled reviews on request of the study team at a demand and frequency determined by the severity of reported adverse events.

The DSMC will be supplied with a safety report at the end of the study, in the event of an SAE, or if requested at any time by the CI or DSMC members.

The Chair of the DSMC will also be contacted for advice where the CI feels independent advice or review is required.

ELIGIBILITY:
Inclusion Criteria:

* Resident near LSTM (<1hr drive) for the duration of the study period
* Allows the investigators to discuss the volunteer's medical history with their GP
* Females of childbearing potential with a negative urine pregnancy test at screening and willing to practice adequate birth control measures during the study.
* Fluent spoken English - to ensure a comprehensive understanding of the research project and their proposed involvement
* Capacity to provide written informed consent
* Able and willing (in the investigators opinion) to comply with all the study requirements

Exclusion Criteria:

* Laboratory evidence at screening of latent M. tb infection as indicated by a positive ELISPOT response to ESAT6 or CFP10 antigens
* Clinical, radiological, or laboratory evidence of current active TB disease
* Previous vaccination with BCG, or any candidate TB vaccine
* Within the last year had close household contact with an individual with smear positive pulmonary tuberculosis
* Clinically significant history of skin disorder, allergy, immunodeficiency (including HIV), cancer, cardiovascular disease, respiratory disease, gastrointestinal disease, liver disease, renal disease, endocrine disorder, neurological illness or psychiatric disorder.
* Current medical issues

  * Acute respiratory tract infection in the four weeks preceding recruitment
  * Any uncontrolled medical or surgical condition at the discretion of the study doctor
* Maternal

  * Female participants who are pregnant
  * Female participants who are lactating
  * Female participants who intend to become pregnant during the study
  * Female participants who are unable to take contraception measures during the study
* Smoking

  * Current (defined as ≥5/week) or ex-smoker (cigarettes / cigars / e-cigarette / vaping / smoking of recreational drugs) in the last 6 months.
  * Previous significant smoking history (more than 20 cigarettes per day for 20 years or the equivalent [>20 pack years]).
* Current alcohol and recreational drug use

  * Regularly drinks ≥3units/day (male) or ≥2units/day (female)
  * Uses recreational drugs
  * Participants may be excluded at the discretion of the research clinician
* Concurrent oral or systemic steroid medication or the concurrent use of other immunosuppressive agents
* History of anaphylaxis to vaccination or any allergy likely to be exacerbated by any component of the challenge agent
* Has received any vaccination within one month of screening visit.
* Has not completed at least two COVID-19 vaccination doses
* Any abnormality of screening blood or urine tests that is deemed to be clinically significant or that may compromise the safety of the volunteer in the study b
* Positive HBsAg, HCV or HIV antibodies
* Current involvement in another trial that involves regular blood tests or an investigational medicinal product
* Use of an investigational medicinal product or non-registered drug, live vaccine, or investigational medical device for four weeks prior to dosing with the study challenge agent
* Administration of immunoglobulins and/or any blood products within the three months preceding the planned challenge date
* Participants who meet STOP criteria at the time of screening (see table 2)
* Any other issue which, in the opinion of the study staff, may

  * Put the participant or their contacts at risk because of participation in the study,
  * Adversely affect the interpretation of the study results, or
  * Impair the participant's ability to participate in the study.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-03-01 (Estimated)

PRIMARY OUTCOMES:
To quantify BCG recovered from the intradermal BCG challenge site. | Day 14 (post BCG injection), phase A.
  Culture and PCR quantification of BCG at intradermal challenge site by punch biopsy at day 14, Phase A.

SECONDARY OUTCOMES:
To monitor for adverse events and any serious adverse events in participants | Daily symptom diary for 14 days, clinic review on day 2, 7, 14, 21 and 28 post BCG injection
  Actively (solicited) and passively collected data on adverse events.
Confirm agreement between BCG recovery between punch biopsy and minimally invasive skin biopsy. | Day 14, phase A.
  Pairwise comparison between culture and PCR quantification by punch and micro skin biopsy.
Confirm agreement between BCG recovery between punch biopsy and minimally invasive skin scrape. | Day 14, phase A.
  Pairwise comparison between culture and PCR quantification by punch biopsy and skin scrape.
Longitudinal quantification of BCG recovery from the intradermal BCG challenge site. | Day 2, 7, 14, 21, 28, Phase B
  Culture and PCR quantification of BCG at intradermal challenge site by non-invasive skin swab/skin scrape/ skin microbiopsy.
Evaluate the immune response to BCG at intradermal injection site from skin biopsy | Day 2, 7, 14, 21, 28, Phase B.
  Microbiopsy cell pellet examined for immune cell differentiation using single cell flow cytometry
Assess cellular immune response to BCG in systemic circulation. | Day 2, 7, 14, 21, 28, Phase B.
  Ex Vivo Interferon γ (IFN-γ) Enzyme-Linked Immunospot (ELISpot) assays will be performed on freshly isolated PBMCs from all participants. Results will be reported as spot-forming cells per million PBMCs.
Measure antibody response to BCG injection in respiratory mucosa. | Day 2, 7, 14, 21, 28, Phase B.
  Nasosorption samples analysed for antibody response to BCG using standard enzyme-linked immunosorbent assays (ELISA)
Measure cellular immune response to BCG injection in respiratory mucosa. | Day 2, 7, 14, 21, 28, Phase B.
  Nasal scrape pellet examined for immune cell differentiation using single cell flow cytometry
Assess antibody response to BCG injection in systemic circulation | Day 2, 7, 14, 21, 28, Phase B.
  Serum samples analysed for antibody response to BCG using standard enzyme-linked immunosorbent assays (ELISA)

CONTACTS AND LOCATIONS:
Overall Officials: Ben Morton, MD. MPH, MBChB, Principal Investigator — Liverpool School of Tropical Medicine
Locations (1):
- Liverpool School of Tropical Medicine, Liverpool, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Data may be shared on suitable direct request from individual researchers to the chief investigator.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: At the end of study
Access Criteria: Data may be shared on suitable direct request from individual researchers to the chief investigator.

REFERENCES:
- [Background] Minassian AM, Ronan EO, Poyntz H, Hill AV, McShane H. Preclinical development of an in vivo BCG challenge model for testing candidate TB vaccine efficacy. PLoS One. 2011;6(5):e19840. doi: 10.1371/journal.pone.0019840. Epub 2011 May 24. PMID 21629699
- [Background] Minassian AM, Satti I, Poulton ID, Meyer J, Hill AV, McShane H. A human challenge model for Mycobacterium tuberculosis using Mycobacterium bovis bacille Calmette-Guerin. J Infect Dis. 2012 Apr 1;205(7):1035-42. doi: 10.1093/infdis/jis012. PMID 22396610
- [Background] Harris SA, Meyer J, Satti I, Marsay L, Poulton ID, Tanner R, Minassian AM, Fletcher HA, McShane H. Evaluation of a human BCG challenge model to assess antimycobacterial immunity induced by BCG and a candidate tuberculosis vaccine, MVA85A, alone and in combination. J Infect Dis. 2014 Apr 15;209(8):1259-68. doi: 10.1093/infdis/jit647. Epub 2013 Nov 23. PMID 24273174
- [Derived] Carter E, Morton B, ElSafadi D, Jambo K, Kenny-Nyazika T, Hyder-Wright A, Chiwala G, Chikaonda T, Chirwa AE, Gonzalez Sanchez J, Yip V, Biagini G, Pennington SH, Saunderson P, Farrar M, Myerscough C, Collins AM, Gordon SB, Ferreira DM. A feasibility study of controlled human infection with intradermal Bacillus Calmette-Guerin (BCG) injection: Pilot BCG controlled human infection model. Wellcome Open Res. 2024 Jun 5;8:424. doi: 10.12688/wellcomeopenres.19811.2. eCollection 2023. PMID 39219857